CLINICAL TRIAL: NCT06408246
Title: ACE-D: Accelerating Cognition-guided Signatures to Enhance Translation in Depression: Clinical Trial
Acronym: ACE-D
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Leanne Williams, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 75568
Record Dates: First submitted 2024-05-06; First posted 2024-05-10 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Guanfacine; Sertraline

STUDY DESIGN:
Intervention Model Description: Participants in C+ and C- subgroups will be randomized to one of two treatment arms
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sertraline + Guanfacine (Experimental): We will conduct a parallel-group, double-blind randomized trial at Stanford Bay Area and Chicago sites, identifying 160 participants with a prominent clinical cognitive signature (C+) and relative absence of the signature (C-). We will enrich for C+, the signature of interest, at a 2:1 ratio. Participants will be randomly assigned to receive guanfacine (shown to ameliorate cognitive control deficits in our preliminary data) plus sertraline or placebo plus sertraline.
  Interventions: Drug: Guanfacine
- Sertraline + Placebo (Experimental): We will conduct a parallel-group, double-blind randomized trial at Stanford Bay Area and Chicago sites, identifying 160 participants with a prominent clinical cognitive signature (C+) and relative absence of the signature (C-). We will enrich for C+, the signature of interest, at a 2:1 ratio. Participants will be randomly assigned to receive guanfacine (shown to ameliorate cognitive control deficits in our preliminary data) plus sertraline or placebo plus sertraline.
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Guanfacine — Guanfacine immediate release is an established and safe FDA-approved treatment that acts directly by stimulating α2A adrenoceptors.
  Arms: Sertraline + Guanfacine
Drug: Sertraline — Sertraline is a well-tolerated FDA-approved antidepressant that is among the most widely prescribed medications for depression.
  Arms: Sertraline + Placebo

SUMMARY:
The purpose of this study is to understand how a psychotropic medication called guanfacine affects brain network functioning in humans, and how this function interacts with cognitive impairments in people experiencing depressive symptoms.

DETAILED DESCRIPTION:
The investigators will conduct a parallel-group, double-blind randomized trial at Stanford Bay Area and Chicago sites, identifying 160 participants across Stanford University and the University of Illinois Chicago with a prominent clinical cognitive signature (C+) and relative absence of the signature (C-).

If you are eligible and choose to participate based off of your answers on the screening survey, the investigators will call you on the number you have provided to verify participants' responses and answer any additional questions you may have about the study.

The first screening visit will consist of obtaining participants' informed consent to participate in the study, completing cognitive testing, answering questions about participants' thoughts and feelings, and providing information about participants' medical and psychiatric history. In addition, this initial screening visit will consist of undergoing an EKG with a medical professional.

If participants are deemed eligible at this phase, the investigators will ask participants to come in for another in-person visit (3 hours) that would involve a non-invasive brain scan. If a participant Is eligible, they will be randomized to receive guanfacine plus sertraline or placebo plus sertraline for an 8 week treatment phase.

Starting week 1 and for every other week during the 8-week treatment phase, participants will complete surveys, passive sampling with the BiAffect application, and conduct cognitive testing. Additionally, starting week 2 and every other week thereafter, participants will conduct a virtual or in-person physician visit. At the end of week 8, the investigators will conduct an MRI visit that resembles the initial MRI visit. Participants will be unblinded over weeks 9-10 to arrange for the participants transition out of the trial.

ELIGIBILITY:
Inclusion Criteria

* 18-60 years of age
* Meets DSM-5-TR diagnostic criteria for current, past, or recurrent nonpsychotic MDD established via the participant's medical record and confirmed with using the Mini International Neuropsychiatric Interview (MINI Plus) when the diagnosis is not clear in the medical record
* At least moderately severe depression as defined as a score of 10 or higher on the PHQ-9
* Meets criteria for cognitive impairment (<=-.5 standard deviation below healthy norms) or intact cognition (within healthy range) subgroups based on a computerized behavioral tests of cognitive control performance (WebNeuro) relative to healthy norms
* Usual treating physician support for participation in the study (including that patients currently on psychotropics who can be safely tapered may be tapered off to participate but must wait at least 5 half-lives prior to first scan);
* Fluent and literate in English; and g) written informed consent.

Exclusion Criteria.

* Suicidal ideations representing imminent risk, defined by a score of ≥ 8 on the MINI Plus, or by clinician judgement
* History of a DSM-5 bipolar disorder (I, II, not otherwise specified) or psychosis (current or lifetime) established via the participant's medical record and confirmed using the MINI Plus as necessary
* History of DSM-5 alcohol or substance use disorder in the last 6 months established via the participant's medical record and confirmed using the MINI Plus as necessary
* Current DSM-5 PTSD, OCD, ADHD, and/or ED established via the participant's medical record and confirmed using the MINI Plus as necessary
* Current or lifetime history of medical illness or brain injury that may interfere with assessments
* Severe impediment to vision, hearing, and/or hand movement, likely to interfere with protocols
* Pregnant, breastfeeding, or unwilling or unable to use adequate birth control throughout the study
* 3.0T MRI scanner contraindications
* Concurrent participation in other intervention studies
* Current use of psychotropic medications contraindicated by GIR or the standard antidepressant medication, sertraline, to which subjects could be randomized
* Prior inadequate response sertraline or guanfacine
* General medical condition or disorder that is deemed by study physicians to be unsafe for GIR as reported by patient or found on medical screening (i.e., kidney or liver impairment, hypotension as defined by SBP ≤ 90 and/or DBP ≤ 60 and/or bradycardia as defined by HR ≤ 55 on 2 of 3 separate measurements at least 5 minutes apart, history of syncope, EKG abnormalities, or family history of cardiac events)
* Positive drug screen for any substance deemed by the study physician to be unsafe for use with GIR in combination with other screening information
* Current use of a strong CYP3A4 inhibitor or inducer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Remission of depressive symptoms | 8 weeks
  A score of <=5 on the PHQ-9

SECONDARY OUTCOMES:
Change in disability | 8 weeks
  Score on the Sheehan Disability Scale which ranges from 0 to 30
Change in quality of Life | 8 weeks
  Score on the Short Form 8 Health Survey (SF-8) which ranges from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Williams, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford Psychiatry and Behavioral Sciences Department, Palo Alto, California
  - University of Illinois at Chicago, Chicago, Illinois